CLINICAL TRIAL: NCT02370238
Title: A Randomized, Double-blind, Placebo-controlled Phase 2 Study of Paclitaxel in Combination With Reparixin Compared to Paclitaxel Alone as Front-line Therapy for Metastatic Triple- Negative Breast Cancer (FRIDA)
Brief Title: A Double-blind Study of Paclitaxel in Combination With Reparixin or Placebo for Metastatic Triple-Negative Breast Cancer
Acronym: FRIDA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REP0114; 2014-004796-23 (EudraCT Number)
Record Dates: First submitted 2015-02-11; First posted 2015-02-24 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Breast Cancer
Keywords: Triple negative metastatic breast cancer; Cancer Stem Cells
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; reparixin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- paclitaxel+reparixin (Experimental): paclitaxel 80 mg/m2 i.v. (Days 1, 8, and 15) + reparixin oral tablets 1200 mg t.i.d.
  continuing from D 1 to Day 21 of 28-day cycle
  Interventions: Drug: paclitaxel; Drug: Reparixin
- paclitaxel+placebo (Active Comparator): paclitaxel 80 mg/m2 i.v. (Days 1, 8, and 15) + placebo oral tablets 1200 mg t.i.d. continuing from D 1 to Day 21 of 28-day cycle
  Interventions: Drug: paclitaxel; Drug: placebo

INTERVENTIONS:
Drug: paclitaxel — paclitaxel 80 mg/m2 i.v. (Days 1, 8, and 15)
Drug: Reparixin — reparixin oral tablets 1200 mg t.i.d. continuing from D 1 to Day 21 of 28-day cycle
  Other Names: REP
  Arms: paclitaxel+reparixin
Drug: placebo — placebo oral tablets 1200 mg t.i.d. continuing from D 1 to Day 21 of 28-day cycle
  Arms: paclitaxel+placebo

SUMMARY:
The Objectives of this study:

The primary objective of the study was to evaluate progression-free survival (PFS) (defined as the number of days between the date of randomization and the date of clinical disease progression (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1, as assessed by Independent Radiology Review, or death for any cause, whichever occured first) in patients with metastatic triple-negative breast cancer (TNBC) treated with the combination of paclitaxel and orally administered reparixin compared to paclitaxel alone.

The secondary objectives were:

* To determine overall survival (OS).
* To evaluate objective response rates (ORR).
* To determine median PFS (mPFS).
* To assess the safety of the combination of paclitaxel and orally administered reparixin (referred to as combination treatment).

DETAILED DESCRIPTION:
The study is a two arm, phase 2 study to evaluate the efficacy of the combination of paclitaxel and reparixin compared to paclitaxel and placebo in metastatic TNBC patients.

In the study two groups There were two groups:

Group 1: paclitaxel 80 mg/m2 intravenous (i.v.) (Days 1, 8, and 15 of 28-day cycle) + reparixin oral tablets 1200 mg three times a day (t.i.d.) continuing from Day 1 to Day 21.

Group 2: paclitaxel 80 mg/m2 i.v. (Days 1, 8, and 15 of 28-day cycle) + placebo oral tablets 1200 mg t.i.d. continuing from Day 1 to Day 21.

Study drug (reparixin/placebo) was administered with water prior to the start of the i.v. paclitaxel infusion on Cycle 1, Day 1 and then administered approximately every eight hours (six to ten hours) for 21 consecutive days during each cycle with seven days off-treatment between each cycle. It was preferable that reparixin was taken with food. However, if the patient was unable to eat, study drug was allowed to be administered. When in combination with paclitaxel (Day 1, 8 and 15 of each cycle), reparixin or placebo was administered every approximately eight hours with about 250 mL water and a light meal or snack. Paclitaxel was administered in combination with study drug (reparixin/placebo) as an i.v. infusion on Days 1, 8 and 15 of each 28-day cycle.

On Cycle 1, Day 1, paclitaxel was administered at the clinic after the administration of study drug (reparixin/placebo). From that point forward, study drug (reparixin/placebo) was self-administered t.i.d. for 21 days. Combination treatment (three weeks on and one week off) continued until PD according to RECIST criteria version 1.1, withdrawal of consent or unacceptable toxicity, whichever occurred first.

The next clinic visits were on Days 8 and 15 when a paclitaxel infusion was administered to the patient. The patients returned to the clinic again on Day 29/Day 1 of the next cycle.

Tumor response and/or progression assessments were performed and documented every eight weeks according to RECIST criteria version 1.1. Metastatic tissue samples were analyzed for evaluation of CD24-CD44+ and aldehyde dehydrogenase positive (ALDH+) CSCs.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged ≥ 18 years.
2. Patients with pathologically documented metastatic triple negative breast cancer (TNBC), eligible for treatment with paclitaxel. Paraffin-embedded tissue must be available from metastatic sites, if reasonably accessible, or from the primary tumor, to confirm the diagnosis of TNBC and for correlative studies (only on metastatic tissue). Fifteen slides can be obtained if the full block is not available to be sent or released.

   TNBC will be defined as breast cancer with <1% ER+ and <1% PgR+ cells, and HER2 immunohistochemistry score of 0 or 1+ and/or in situ hybridization (ISH) with HER2 gene copy number <4 or a ratio of less than 2 between HER2 gene copy number and centromere of chromosome 17. Patients whose metastatic disease is TNBC are eligible even when their primary tumor expressed hormone receptors and/or HER2.
3. Patients must be newly diagnosed metastatic or must have relapsed following a prior (neo)adjuvant chemotherapy regimen. If a taxane (i.e., paclitaxel or docetaxel) was administered as part of the (neo)adjuvant regimen, PD must have occurred > 12 months from the end of previous (neo)adjuvant treatment. For non-taxane (neo)adjuvant regimen, PD must have occurred > 6 months from the end of previous (neo)adjuvant treatment
4. Patients with at least one baseline measurable lesion according to RECIST criteria version 1.1.
5. Zubrod (Eastern Co-operative Oncology Group [ECOG]) Performance Status (PS) of 0-1.
6. Life expectancy of at least three months.
7. Patients must be able to swallow and retain oral medication (intact tablet).
8. Able to undergo all screening assessments outlined in the protocol.
9. Adequate organ function (defined by the following parameters):

   1. Serum creatinine < 140 μmol/L (< 1.6 mg/dL) or creatinine clearance > 60 mL/min.
   2. Serum hemoglobin ≥ 9 g/dL; absolute neutrophil count ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L.
   3. Serum bilirubin ≤ 1.5 x upper normal limit (UNL) except patients with Gilbert's syndrome
   4. Serum alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5 x UNL but ≤ 5.0 x UNL in case of liver metastases; alkaline phosphatase (ALP) ≤ UNL but i) ≤ 2.5 x UNL in case of liver metastases and ii) ≤ 5 UNL in case of bone metastases; albumin ≥ 2.5 g/dl.
10. No history or evidence by CT scan or MRI, of brain metastases or leptomeningeal disease.
11. No known hepatitis B virus (not due to immunization), hepatitis C virus, human immunodeficiency virus-I and -II positive status.
12. Dated and signed IEC/IRB-approved informed consent.

Exclusion Criteria:

1. Prior therapy for metastatic TNBC (chemotherapy, hormone therapy or biological therapy), Patients may receive bisphosphonates and other therapies to treat bone metastases, however if used, bone lesions will not be considered as measurable disease.
2. Less than four weeks since last radiotherapy (excluding palliative radiotherapy).
3. Pregnancy or lactation or unwillingness to use adequate method of birth control.
4. Neurological or psychiatric disorders which may influence understanding of study and informed consent procedures.
5. Active or uncontrolled infection.
6. Malabsorption syndrome, disease significantly affecting gastrointestinal function.
7. G>1 pre-existing peripheral neuropathy
8. Any other invasive malignancy from which the patient has been disease-free for less than 5 years with the exception of curatively treated basal or squamous cell skin cancer
9. Hypersensitivity to:

   1. paclitaxel
   2. ibuprofen or to more than one non-steroidal anti-inflammatory drug.
   3. medications belonging to the class of sulfonamides, with the exception of sulfanilamides (e.g., sulfamethoxazole).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori J Goldstein, MD, Principal Investigator — FASCOFox Chase Cancer Center
Locations (77):
- United States (32):
  - Southern Cancer Center, Mobile, Alabama
  - CBCC Global Research a Comprehensive Blood and Cancer Center, Bakersfield, California
  - Florida Cancer Specialists, Daytona Beach, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Atlanta Cancer Care, Alpharetta, Georgia
  - Northside Hospital, Inc.-Georgia Cancer Specialists, Athens, Georgia
  - Atlanta Cancer Care, Atlanta, Georgia
  - Northside Hospital, Inc., Atlanta, Georgia
  - Northside Hospital, Inc.-Georgia Cancer Specialists, Canton, Georgia
  - Atlanta Cancer Care, Conyers, Georgia
  - Atlanta Cancer Care, Cumming, Georgia
  - Atlanta Cancer Care, Decatur, Georgia
  - Northside Hospital, Inc.-Georgia Cancer Specialists, Decatur, Georgia
  - Atlanta Cancer Care, Jonesboro, Georgia
  - Northside Hospital, Inc.-Georgia Cancer Specialists, Macon, Georgia
  - Northside Hospital, Inc.-Georgia Cancer Specialists, Marietta, Georgia
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Northside Hospital, Inc.-Georgia Cancer Specialists, Sandy Springs, Georgia
  - Swedish Covenant, Chicago, Illinois
  - Mid Illinois Hematology & Oncology Associates, Ltd., Normal, Illinois
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Summit Medical Group, Morristown, New Jersey
  - Regional Cancer Care Associates, Sparta, New Jersey
  - Waverly Hematology Oncology, Cary, North Carolina
  - Hematology and Oncology Associates of Northeast PA, Dunmore, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology PLLC, Chattanooga, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Overlake Medical Center, Bellevue, Washington
  - Fox Valley Hematology and Oncology, SC, Appleton, Wisconsin
- Belgium (5):
  - Algemeen Ziekenhuis Klina, Brasschaat
  - Cliniques Universitaires Saint- LUC UCL, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - CHU Ambroise Paré, Mons
  - AZ St Elisabeth, Namur
- Czechia (7):
  - Masaryk Memorial Cancer Institute, Brno
  - Nemocnice Horovice a.s., Hořovice
  - Fakultni nemocnice Hradec Králové, Hradec Králové
  - Fakultní nemocnice Královské Vinohrady, Prague
  - Onkologická klinika VFN a 1.LF UK, Prague
  - Fakultní nemocnice v Motole, Onkologická klinika 2. LF UK a FN Motol, Prague
  - Krajská nemocnice T.Bati, a. s., Zlín
- France (8):
  - Centre Paul Papin, Angers
  - Centre François Baclesse, Caen
  - Centre hospitalier de Saint-Brieuc, Yves Le Foll, La Roche-sur-Yon
  - Centre Hospitalier Universitaire (CHU) De Limoges - Hopital Dupuytren, Limoges
  - Institut Paoli Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Hôpital Européen Georges Pompidou, Paris
  - Medicale Centre René Gauducheau, Saint-Herblain
- Italy (12):
  - Ospedale "Di Summa-Perrino", Brindisi
  - Azienda Ospedaliero-Universitaria, Cagliari
  - Azienda Ospedaliero - Universitaria, Policlinico Vittorio Emanuele, Catania
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Ospedale dell'Angelo, Mestre
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera, Ospedale San Carlo Borromeo, Milan
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro
  - Nuovo Ospedale, Prato
  - Azienda Opspedaliero Universitaria Santa Maria della Misericordia, Udine
  - Ospedale SS Giovanni e Paolo, Venezia
- Poland (6):
  - Bialostockie Centrum Onkologii im. Marii Sklodowskiej - Curie, Bialystok
  - Wojewódzkie Centrum Onkologii, Gdansk
  - Centrum Onkologii Ziemi Lubelskiej im. sw. Jana z Dukli, Lublin
  - Uniwersytet Medyczny im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Mrukmed. Lekarz Beata Madej Mruk i Partner. Spólka Partnerska Oddzial nr 1 w Rzeszowie, Rzeszów
  - Magodent Sp. z o. o., Warsaw
- Spain (7):
  - Centro Oncológico Regional de Galicia, Servicio de Oncologia Medica, A Coruña, Galicia
  - Complejo Hospitalario Universitario La Coruña, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Centro Integral Oncológico Clara Campal, Hospital de Madrid Norte-San Chinarro, Madrid
  - C. Hospital Xeral-Cies, Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gong YT, Zhang LJ, Liu YC, Tang M, Lin JY, Chen XY, Chen YX, Yan Y, Zhang WD, Jin JM, Luan X. Neutrophils as potential therapeutic targets for breast cancer. Pharmacol Res. 2023 Dec;198:106996. doi: 10.1016/j.phrs.2023.106996. Epub 2023 Nov 14. PMID 37972723
- [Derived] Schott AF, Goldstein LJ, Cristofanilli M, Ruffini PA, McCanna S, Reuben JM, Perez RP, Kato G, Wicha M. Phase Ib Pilot Study to Evaluate Reparixin in Combination with Weekly Paclitaxel in Patients with HER-2-Negative Metastatic Breast Cancer. Clin Cancer Res. 2017 Sep 15;23(18):5358-5365. doi: 10.1158/1078-0432.CCR-16-2748. Epub 2017 May 24. PMID 28539464
- See also: Corporate webpage — http://www.dompe.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 194 enrolled patients, 123 were randomized and included in the ITT Population: 62 patients in Group 1 and 61 patients in Group 2.
Pre-assignment Details: Due to extreme enrollment difficulties during the first 6 months of 2018, enrollment to the study was terminated early (30 July 2018) and the final sample size is equal to 123 randomized patients.
Groups:
- Paclitaxel+Reparixin (Group 1): paclitaxel 80 mg/m2 i.v. (Days 1, 8, and 15) + reparixin oral tablets 1200 mg t.i.d. continuing from D 1 to Day 21 of 28-day cycle.
  Duration of Treatment: 28-day cycles of combination therapy reparixin oral tablets + paclitaxel intravenous weekly three weeks on and one week off until disease progression according to RECIST criteria version 1.1, withdrawal of consent or unacceptable toxicity, whichever occurred first.
- Paclitaxel+Placebo (Group 2): paclitaxel 80 mg/m2 i.v. (Days 1, 8, and 15) + placebo oral tablets 1200 mg t.i.d. continuing from D 1 to Day 21 of 28-day cycle.
  Duration of Treatment: 28-day cycles of combination therapy placebo oral tablets + paclitaxel intravenous weekly three weeks on and one week off until PD according to RECIST criteria version 1.1, withdrawal of consent or unacceptable toxicity, whichever occurred first.
Period: Overall Study
Arm/Group | Paclitaxel+Reparixin (Group 1) | Paclitaxel+Placebo (Group 2)
Started | 62 | 61
ITT Population | 62 | 61
Safety Population | 61 | 60
Responsable-evaluable Population | 57 | 54
Completed | 15 | 16
Not Completed | 47 | 45
Not completed — Death | 42 | 35
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population consisted of 121 patients who took at least one dose of study treatment
Groups:
- Paclitaxel+Reparixin (Group 1) - Safety Population: paclitaxel 80 mg/m2 i.v. (Days 1, 8, and 15) + reparixin oral tablets 1200 mg t.i.d. continuing from D 1 to Day 21 of 28-day cycle.
  Duration of Treatment: 28-day cycles of combination therapy reparixin oral tablets + paclitaxel intravenous weekly three weeks on and one week off until disease progression according to RECIST criteria version 1.1, withdrawal of consent or unacceptable toxicity, whichever occurred first.
- Paclitaxel+Placebo (Group 2) - Safety Population: paclitaxel 80 mg/m2 i.v. (Days 1, 8, and 15) + placebo oral tablets 1200 mg t.i.d. continuing from D 1 to Day 21 of 28-day cycle.
  Duration of Treatment: 28-day cycles of combination therapy placebo oral tablets + paclitaxel intravenous weekly three weeks on and one week off until PD according to RECIST criteria version 1.1, withdrawal of consent or unacceptable toxicity, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Paclitaxel+Reparixin (Group 1) - Safety Population | Paclitaxel+Placebo (Group 2) - Safety Population | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 44 | 88
  >=65 years | 17 | 16 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 60 | 121
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 48 | 54 | 102
  Unknown or Not Reported | 10 | 4 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 45 | 49 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 4 | 14
Region of Enrollment [Number; unit: participants]
  Belgium | 4 | 6 | 10
  United States | 15 | 19 | 34
  Czechia | 3 | 8 | 11
  Poland | 6 | 3 | 9
  Italy | 16 | 12 | 28
  France | 10 | 4 | 14
  Spain | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the number of days between the date of randomization and the date of clinical disease progression, according to RECIST criteria version 1.1, as assessed by Independent Radiology Review, or to death due to any cause, whichever occurred first.
  Patients must have completed at least one course of treatment and performed at least one disease assessment to be considered evaluable for response.
Time Frame: Baseline up to every 8 weeks until disease progression or death, whichever occurs first, up to 721 days
Population: The Intent-to-Treat (ITT) Population consisted of all patients who are randomized and was based upon the randomized treatment, regardless of the treatment actually received. Patients were in the ITT analysis whether or not they received study drug. The primary and secondary efficacy analyses were presented primarily for the ITT Population.
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Paclitaxel+Reparixin (Group 1) - ITT Population: paclitaxel 80 mg/m2 i.v. (Days 1, 8, and 15) + reparixin oral tablets 1200 mg t.i.d. continuing from D 1 to Day 21 of 28-day cycle.
  Duration of Treatment: 28-day cycles of combination therapy reparixin oral tablets + paclitaxel intravenous weekly three weeks on and one week off until disease progression according to RECIST criteria version 1.1, withdrawal of consent or unacceptable toxicity, whichever occurred first.
Arm/Group | Paclitaxel+Reparixin (Group 1) - ITT Population | Paclitaxel+Placebo (Group 2)
Number analyzed (Participants) | 62 | 61
Days | 166 [62 to 292] | 171 [105 to 393]
Statistical Analysis 1: Comparison: Paclitaxel+Reparixin (Group 1) - ITT Population vs Paclitaxel+Placebo (Group 2); Test type: Superiority; p = 0.589, Log Rank — p-value based on a log-rank test stratified by randomized sub-populations, newly diagnosed metastatic patients and patients that had relapsed following a prior (neo)adjuvant chemotherapy regimen; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.71 to 1.81]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization until death due to any cause. For patients who did not die, time of death was censored at the date of last contact.
  Patients must have completed at least one course of treatment and performed at least one disease assessment to be considered evaluable for response.
Time Frame: Baseline until death due to any cause, up to 985 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Paclitaxel+Reparixin (Group 1) - ITT Population | Paclitaxel+Placebo (Group 2)
Number analyzed (Participants) | 62 | 61
Days | 483 [272 to 812] | 531 [334 to 787]
Statistical Analysis 1: Comparison: Paclitaxel+Reparixin (Group 1) - ITT Population vs Paclitaxel+Placebo (Group 2); Test type: Superiority; p = 0.897, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.64 to 1.65]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of patients achieving CR or PR in the Evaluable Population. The response rate was calculated from the independently reviewed assessment best response. In case of PR or CR, only confirmed cases were considered to be responses.
  Complete Response (CR) = Disappearance of all target lesions; Partial Response (PR) = >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Patients with unknown or missing response, including response of "not all evaluated" or "unable to determine", were treated as non-responders; i.e., they were included in the denominator when calculating the percentages.
  Patients must have completed at least one course of treatment and performed at least one disease assessment to be considered evaluable for response.
Time Frame: Baseline up to every 8 weeks until documented disease progression, up to 56 months
Population: Responsible-evaluable population: this population consisted of all patients who had completed at least one cycle of treatment and had a baseline assessment and have undergone at least one post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Paclitaxel+Reparixin (Group 1) - ITT Population | Paclitaxel+Placebo (Group 2)
Number analyzed (Participants) | 57 | 54
Percentage of patients | 28.1 [17.0 to 41.5] | 25.9 [15.0 to 39.7]
Statistical Analysis 1: Comparison: Paclitaxel+Reparixin (Group 1) - ITT Population vs Paclitaxel+Placebo (Group 2); Test type: Superiority; p = 0.667, Zelen's test — P-value is based on Zelen's test for homogeneity of the odds ratios; Odds Ratio (OR) = 1.262, 95% CI 2-sided [0.4909 to 3.963]

4. Secondary Outcome: Median Progression-free Survival (mPFS)
Description: PFS was defined as the time from randomization to first documentation of disease progression, according to RECIST criteria version 1.1, as assessed by Independent Radiology Review, or to death due to any cause, whichever occurred first. For each treatment group, the Kaplan-Meier estimates for the median PFS time, the first and third quartiles were presented, along with approximate 95% confidence intervals if there were a sufficient number of progressions or deaths.
  Patients must have completed at least one course of treatment and performed at least one disease assessment to be considered evaluable for response.
Time Frame: At screening and every 8 weeks, up to 721 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Paclitaxel+Reparixin (Group 1) - ITT Population | Paclitaxel+Placebo (Group 2)
Number analyzed (Participants) | 62 | 61
Days | 166 [109 to 218] | 171 [117 to 226]

5. Secondary Outcome: Duration of Overall Response (DOR)
Description: Duration of overall response (DOR) in days for the investigator assessments is measured from the time response criteria are first met for CR or PR (whichever is first recorded on the "Disease Response" page on the CRF) until either death or the first date that recurrent or PD is objectively documented (on the "Disease Response" p. on the CRF or the Follow-Up Disease Evaluation page indicates disease progression and there is supporting information in the Disease Status pages) per RECIST version 1.1. Complete Response (CR) = Disappearance of all target lesions; Partial Response (PR) = >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. If a patient is lost to follow-up with no documentation of PD, DOR was censored at the last evaluable tumor assessment. DOR was calculated only for responding patients (PR or CR) as recorded on the CRF page "Disease Response" based upon the RECIST version 1.1.
  Duration of overall response wa
Time Frame: Baseline up to every 8 weeks until documented disease progression, up to 557 days
Population: The Response-Evaluable Population consisted of all patients who had completed at least one cycle of treatment and had a baseline assessment and have undergone at least one post-baseline disease assessment.
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Group 1 - Response Evaluable Population: paclitaxel 80 mg/m2 i.v. (Days 1, 8, and 15) + reparixin oral tablets 1200 mg t.i.d. continuing from D 1 to Day 21 of 28-day cycle.
  Duration of Treatment: 28-day cycles of combination therapy reparixin oral tablets + paclitaxel intravenous weekly three weeks on and one week off until disease progression according to RECIST criteria version 1.1, withdrawal of consent or unacceptable toxicity, whichever occurred first.
- Group 2 - Response-Evaluable Population: paclitaxel 80 mg/m2 i.v. (Days 1, 8, and 15) + placebo oral tablets 1200 mg t.i.d. continuing from D 1 to Day 21 of 28-day cycle.
  Duration of Treatment: 28-day cycles of combination therapy placebo oral tablets + paclitaxel intravenous weekly three weeks on and one week off until PD according to RECIST criteria version 1.1, withdrawal of consent or unacceptable toxicity, whichever occurred first.
Arm/Group | Group 1 - Response Evaluable Population | Group 2 - Response-Evaluable Population
Number analyzed (Participants) | 57 | 54
Days | 293.0 [119.0 to 505.0] | 172.0 [115.0 to 443.0]
Statistical Analysis 1: Comparison: Group 1 - Response Evaluable Population vs Group 2 - Response-Evaluable Population; Test type: Superiority; p = 0.767, Log Rank — For the All Patients group, p-value was based on a log-rank test stratified by actual sub-populations, newly diagnosed metastatic patients and patients that had relapsed following a prior (neo)adjuvant chemotherapy regimen

6. Secondary Outcome: Best Overall Response (BOR)
Description: BOR is defined as the best response among all overall responses (in the order complete response [CR], partial response [PR], stable disease [SD], and progressive disease [PD]) recorded as an independent review response from the start of reparixin or placebo until disease progression/recurrence or end of treatment, or death, whichever comes first. The status of BOR of PR or CR needs to be confirmed by repeat tumor assessment within no less than 4 weeks according to RECIST version 1.1. Complete Response (CR) = Disappearance of all target lesions; Partial Response (PR) = >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. If the status of CR or PR cannot be confirmed by repeat tumor assessment, the best overall response of unconfirmed CR and PR will be PR and SD, respectively. Patients must have completed at least one course of treatment and performed at least one disease assessment to be considered evaluable for response.
Time Frame: From the start of treatment, every 8 weeks, up to 56 months
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Group 1 - Response Evaluable Population | Group 2 - Response-Evaluable Population
Number analyzed (Participants) | 57 | 54
participants
  CR | 1 | 0
  PR | 15 | 14
  SD | 16 | 23
  PD | 22 | 14
  NE | 3 | 3
  Unable to determine | 0 | 0
  Unknown/not done | 0 | 0
Statistical Analysis 1: Comparison: Group 1 - Response Evaluable Population vs Group 2 - Response-Evaluable Population; Test type: Superiority; p = 0.667, Zelen's test — P-value was based on Zelen's test for homogeneity of the odds ratios; Odds Ratio (OR) = 1.101, 95% CI 2-sided [0.437 to 2.790]

7. Secondary Outcome: Number of Treatment-Emergent Adverse Events (TEAEs), Overall and by Grade
Description: Treatment-emergent adverse events (TEAEs) are those which first occur or increase in severity or relationship to study drug after the first dose of study drug and before 30 days after the last dose of study treatment, reparixin/placebo. In the case of missing or partial dates, any AE that could have started on or after first dose date was assumed to be treatment-emergent. In the case of missing or partial dates, imputed dates (see section 10.1 AE date imputation) were used.
Time Frame: Throughout the study, until off-treatment visit (performed 14 to 28 days following the last dose of study drug), up to 985 days
Population: Safety population: this population consisted of all patients who had taken at least one dose of the study treatment and was based upon the treatment they actually received.
Measure: Number; unit: number of events
Arm/Group | Paclitaxel+Reparixin (Group 1) - Safety Population | Paclitaxel+Placebo (Group 2) - Safety Population
Number analyzed (Participants) | 61 | 60
number of events
  Overall | 865 | 730
  Grade 1 (mild) | 563 | 478
  Grade 2 (moderate) | 230 | 194
  Grade 3 (severe) | 67 | 50
  Grade 4 (Life-threatening or disabling) | 2 | 4
  Grade 5 (death) | 3 | 4

8. Secondary Outcome: Serious AEs and Fatal AEs
Description: A serious adverse event (SAE) in human drug trials is defined as any untoward medical occurrence that at any dose
  1. - results in death, (fatal)
  2. - is life-threatening
  3. - requires inpatient hospitalization or causes prolongation of existing hospitalization
  4. - results in persistent or significant disability/incapacity,
  5. - may have caused a congenital anomaly/birth defect, or
  6. - requires intervention to prevent permanent impairment or damage.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Number; unit: number of events
Arm/Group | Paclitaxel+Reparixin (Group 1) - Safety Population | Paclitaxel+Placebo (Group 2) - Safety Population
Number analyzed (Participants) | 61 | 60
number of events
  serious AE | 31 | 25
  Fatal AE | 3 | 4

ADVERSE EVENTS:
Time Frame: Throughout the study, until off-treatment visit (performed 14 to 28 days following the last dose of study drug), up to 985 days.
Description: A Summary of the Most Frequent (i.e., 5 or More Patients Experiencing an Event by Preferred Term in Any Treatment Group) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term is reported.
Arm/Group | Paclitaxel+Reparixin (Group 1) - Safety Population | Paclitaxel+Placebo (Group 2) - Safety Population
All-Cause Mortality (participants affected / at risk) | 42/61 | 35/60
Serious Adverse Events (participants affected / at risk) | 13/61 | 12/60
Other Adverse Events (participants affected / at risk) | 60/61 | 57/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel+Reparixin (Group 1) - Safety Population (N=61) | Paclitaxel+Placebo (Group 2) - Safety Population (N=60)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.92% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel+Reparixin (Group 1) - Safety Population (N=61) | Paclitaxel+Placebo (Group 2) - Safety Population (N=60)
Asthenia (General disorders) | 16 (16) | 13 (13)
Fatigue (General disorders) | 11 (11) | 26 (26)
Pyrexia (General disorders) | 8 (8) | 8 (8)
Oedema peripheral (General disorders) | 7 (7) | 8 (8)
Nausea (Gastrointestinal disorders) | 23 (23) | 22 (22)
Diarrhoea (Gastrointestinal disorders) | 16 (16) | 15 (15)
Constipation (Gastrointestinal disorders) | 14 (14) | 11 (11)
Vomiting (Gastrointestinal disorders) | 9 (9) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 7 (7)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 21 (21) | 21 (21)
Rash (Skin and subcutaneous tissue disorders) | 9 (9) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 13 (13) | 8 (8)
Neuropathy peripheral (Nervous system disorders) | 12 (12) | 11 (11)
Dysgeusia (Nervous system disorders) | 9 (9) | 5 (5)
Dizziness (Nervous system disorders) | 7 (7) | 3 (3)
Paresthesia (Nervous system disorders) | 7 (7) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Urinary tract infection (Infections and infestations) | 6 (6) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 11 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 18 (18) | 8 (8)
Neutropenia (Blood and lymphatic system disorders) | 10 (10) | 7 (7)
Leukopenia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Alanine aminotransferase increased (Investigations) | 8 (8) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 3 (3)
White blood cell count decreased (Investigations) | 3 (3) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 10 (10)
Hot flush (Vascular disorders) | 6 (6) | 6 (6)
insomnia (Psychiatric disorders) | 5 (5) | 4 (4)
Hypertension (Vascular disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT02370238/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT02370238/SAP_001.pdf